CLINICAL TRIAL: NCT02036788
Title: Comparison of Two Tests in the Assessment of the Accuracy of Esophageal Pressure Variations Measurement During Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: Policlinico-11
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Pressure Measurement
Keywords: Esophageal pressure, Mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Postsurgical patients sedated and paralized: Patients admitted to ICU after surgery, treated with mechanical ventilation, sedated and paralized
  Interventions: Other: Thoraco-abdominal compressions
- Postsurgical patients intubated and breathing spontaneously
  Interventions: Other: Occlusion test

INTERVENTIONS:
Other: Occlusion test — Occlusion test to assess the correct positioning of esophageal balloon catheter when the patient is breathing spontaneously.
  Groups: Postsurgical patients intubated and breathing spontaneously
Other: Thoraco-abdominal compressions — Thoraco-abdominal compressions to assess the correct positioning of esophageal balloon catheter when the patient is sedated and paralyzed.
  Groups: Postsurgical patients sedated and paralized

SUMMARY:
Esophageal pressure measurement, obtained with the use of an esophageal balloon catheter, is fundamental to assess mechanical characteristics of the respiratory system during mechanical ventilation. The correct positioning of the catheter (usually at the medium third of the esophagus) is crucial for an accurate measurement of esophageal pressure. Usually the correct positioning of the catheter is verified with an occlusion test (If the patient is breathing spontaneously) or with thoraco-abdominal compressions (if the patient is sedated and paralyzed). Aim of this study is to compare the accuracy of these two methods at different PEEP and esophageal catheter positions.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation for clinical purposes

Exclusion Criteria:

* Hemodynamic instability
* Esophageal diseases
* Refusal of the patient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU after surgery treated with mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Correct esophageal catheter balloon position | 10 minutes after the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Background] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319
- [Background] Hedenstierna G. Esophageal pressure: benefit and limitations. Minerva Anestesiol. 2012 Aug;78(8):959-66. Epub 2012 Jun 14. PMID 22699701
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Higgs BD, Behrakis PK, Bevan DR, Milic-Emili J. Measurement of pleural pressure with esophageal balloon in anesthetized humans. Anesthesiology. 1983 Oct;59(4):340-3. doi: 10.1097/00000542-198310000-00012. PMID 6614543